CLINICAL TRIAL: NCT02686047
Title: Comparing Efficacy and Safety of a Single Intraarticular Injection of a Novel Crosslinked Hyaluronic Acid (HYAJOINT Plus) With Synvisc-One for the Treatment of Knee Osteoarthritis: A Randomized-Controlled, Double-Blind Trial
Brief Title: Comparing One Intraarticular Injection of a Novel HYAJOINT Plus With Synvisc-One for the Treatment of Knee OA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Shu-Fen Sun, MD, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VGHKS14-CT8-12
Record Dates: First submitted 2016-02-11; First posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Hyaluronic acid; Viscosupplementation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the HYAJOINT Plus group (Experimental): the HYAJOINT Plus group received one intraarticular injection of 3 ml HYAJOINT Plus (2% microbial fermented HA, 20 mg/ml).
  Interventions: Device: HYAJOINT Plus
- The Synvisc-One group (Active Comparator): The Synvisc-One group received one injection of 6 ml Synvisc-One (0.8% avian derived HA, 8 mg/ml).
  Interventions: Device: Synvisc-One

INTERVENTIONS:
Device: HYAJOINT Plus — The patients in the HYAJOINT Plus group received one intraarticular injection of 3 ml HYAJOINT Plus (2% microbial fermented HA, 20 mg/ml).
  Other Names: Hyaluronic acid
  Arms: the HYAJOINT Plus group
Device: Synvisc-One — The Synvisc-One group received one injection of 6 ml Synvisc-One (0.8% avian derived HA, 8 mg/ml).
  Arms: The Synvisc-One group

SUMMARY:
Viscosupplementation has been widely used for the treatment of knee osteoarthritis (OA). There is no well controlled trial comparing one injection regimen of HA for the treatment of knee OA. The purpose of this study was to compare the efficacy and safety of one intraarticular injection of a novel crosslinked HA (HYAJOINT Plus) with Synvisc-One for the treatment of knee OA.

DETAILED DESCRIPTION:
In a prospective, randomized controlled, double-blind trial with 6-month follow up, patients with knee OA (Kellgren-Lawrence grade 2 or 3) were randomized to receive one intraarticular injection of 3 ml HYAJOINT Plus (microbial fermented HA, 20 mg/ml) (N=66) or 6 ml Synvisc-One (avian derived HA, 8 mg/ml) (N=66). The primary outcome was change in the visual analog scale (VAS) pain (0-100mm) over 6 months. Secondary outcomes included The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Lequesne index, Timed Up-and-Go test (TUG), single leg stance test (SLS), use of rescue analgesics and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic knee OA with pain for at least 6 months, despite conservative treatment such as analgesics, NSAIDs and/or physical therapy
* average pain on knee movement of 30 mm or greater on a 100-mm VAS

  * grade 2 or 3 knee OA according to the Kellgren-Lawrence grading system based on radiographs taken within the previous 6 months
  * Radiological evidence of bilateral knee OA was accepted if global pain VAS in the contralateral knee was less than 30 mm.

Exclusion Criteria:

* previous orthopedic surgery on the spine or lower limbs
* disabling OA of either hip or foot
* knee instability, clinical apparent joint effusion or marked valgus/varus deformity
* known allergy to avian proteins or HA products
* women ascertained or suspected pregnancy or lactating
* intraarticular injections within the past 6 months
* infections or skin diseases around the target knee
* any specific medical conditions (rheumatoid arthritis, hemiparesis, neoplasm, etc.) that would interfere with the assessments

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
VAS pain score | at 1, 3 and 6 months postinjection
  the change from baseline in the VAS pain score over 6 months.

SECONDARY OUTCOMES:
WOMAC, Likert Scale | at 1, 3 and 6 months postinjection
  a 24-item questionnaire with 3 subscales measuring pain, stiffness, and physical function. Total score is 96 and lower scores indicate better outcomes.
Lequesne index | at 1, 3 and 6 months postinjection
  Maximal score is 24 and higher scores represent worse function.
Timed Up-and-Go test (TUG) | at 1, 3 and 6 months postinjection
  a simple measurement of time in seconds for a person to rise from an armchair, walk 3 meters, turn around, walk back to the chair, and sit down
Single-leg stance test (SLS) | at 1, 3 and 6 months postinjection
  by raising one foot up without touching it to the supported lower extremity with target knee OA and maintain balance for as long as possible.
satisfaction based on a 100 mm VAS | at 1, 3 and 6 months postinjection
  Patients were asked to rate their treatment satisfaction compared to the preinjection condition, based on a 100 mm VAS
The reported adverse events | at 1 week (safety records via phone call), 1, 3 and 6 months after the injection
  based on adverse events reported by the patients during the study period and physical examination findings by the evaluator after injections and at each follow-up visit

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No